CLINICAL TRIAL: NCT07218367
Title: Targeting Infiltrating Glioblastoma Via pH Sensitive Visualization of Tumor and pH Modulation Through Bicarbonate Transporter SLC4A4
Brief Title: Phase I Trial of pH Resections of GBM at VA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCE-002-25S
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: glioblastoma; high grade glioma
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Intervention Model Description: A pH based MRI is carried out, uploaded to intraoperative neuronavigation software, and used in a surgical escalation study to increase amounts of infiltrating pH abnormal tumor removed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pH Resections (Experimental): This is a single arm study so all patients will receive the intervention
  Interventions: Procedure: pH MRI based resection of GBM

INTERVENTIONS:
Procedure: pH MRI based resection of GBM — This will require a chemical exchange saturation transfer MRI followed by surgical resection based on this MRI.

SUMMARY:
Glioblastoma is an infiltrating tumor that is difficult to visualize in surgery and on standard images. A special pH (acid-base) related magnetic resonance imaging (MRI) has been developed to better see infiltrating tumor. In this safety study, the investigators will carry out increased levels of pH based resections of infiltrating tumor to assess the tolerability in VA populations.

DETAILED DESCRIPTION:
Current standard of care therapy and all FDA approved adjuvant therapy for glioblastoma continue to provide less than 12 months of progression free survival (PFS) and less than 24 months of overall survival (OS). There is an extreme need for any novel therapy against glioblastoma that increases progression free survival and overall survival in patients diagnosed with this invasive form of cancer. A significant reason for such a poor prognosis is the infiltrative nature of this tumor in non-enhancing regions (NE) beyond the central contrast-enhancing (CE) portion of tumor, which is difficult to visualize and treat with surgical, medical, or radiotherapeutic means. Since tumor cells exhibit abnormal metabolic behavior leading to extracellular acidification, the investigators theorize a newly developed pH-sensitive MRI technique called amine chemical exchange saturation transfer echoplanar imaging (CEST-EPI) may identify infiltrating NE tumor beyond what is clear on standard MRI with gadolinium contrast. This phase I safety study will use intraoperative CEST-EPI guided resections in glioblastoma at increasing distances from areas of CE tumor to test whether this technique is safe and can remove additional areas of infiltrative NE tumor.

The primary objective of this study is to assess the safety of pH-sensitive amine CEST-EPI guided resections for glioblastoma, with secondary objectives to conduct a preliminary efficacy analysis of these resections in extending progression-free and overall survival and to confirm that resected tissue obtained from pH-sensitive amine CEST-EPI guided resections contain infiltrating NE tumor. If any additional CEST-EPI resection is deemed safe by the safety study, then the recommended maximum resection will be determined, which could potentially lead to improved surgical outcomes and survival for patients with this devastating disease. This novel approach addresses an urgent unmet need in neuro-oncology by potentially enabling more complete tumor resection guided by metabolic activity rather than conventional contrast enhancement patterns.

This is a single center, single arm, phase 1 surgical dose escalation clinical trial with a preliminary efficacy study at the recommended safe maximal resection. Prior to surgery, participants will undergo standard medical clearance and a standard pre-operative MRI with the addition of a pH-weighted amine CEST-EPI MRI scan (adding approximately 15 minutes of scan time). During surgery, tumor specimens will be biopsied for diagnostic confirmation and comparative analysis between standard surgical techniques and CEST-EPI guided resection. The study will follow a rule-based approach for resection escalation (based on an i3+3 design) with increasing distances from contrast enhancing tumor (0.7 cm, 1.4 cm, 2.1 cm, or 2.8 cm). Safety will be assessed by monitoring for pre-defined resection limiting toxicities (RLTs) during the post-operative period, with follow-up MRIs at 24 hours, 2 weeks, and 4 weeks post-surgery. Based on safety data, a maximum tolerated resection will be determined, and if found safe, a preliminary efficacy study comparing to historical controls may be conducted. Participants will receive standard post-operative care and adjuvant therapy per established guidelines for glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Karnofsky Performance Scale (KPS) of 70 or higher
* Suspected, newly diagnosed or recurrent IDH wild type WHO IV glioblastoma presenting as an intra-axial
* Expansile contrast-enhancing mass without evidence of metastatic disease

Exclusion Criteria:

* Diagnostic uncertainty such as history of extracranial malignancy or autoimmune disease
* Medical conditions prohibiting anesthesia or surgery
* Tumors involving eloquent brain areas as defined by MRI signal
* primary motor cortex, primary sensory cortex, sensorimotor fibers, primary language areas, arcuate fasciculus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Resection related adverse events | 1 month
  Safety as described by surgical complication rates by the data safety and monitoring board

CONTACTS AND LOCATIONS:
Overall Officials: Kunal S Patel, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No